CLINICAL TRIAL: NCT06632379
Title: AtorvaStatin Postpartum and Reduction of Cardiovascular risK (SPARK): A Randomized Placebo-controlled Trial of Atorvastatin Postpartum for Reduction of Cardiovascular Risk
Brief Title: AtorvaStatin Postpartum and Reduction of Cardiovascular risK
Acronym: SPARK
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Tracy Caroline Bank, MD (Fellow), Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024H0320
Record Dates: First submitted 2024-09-24; First posted 2024-10-09 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Hypertensive Disorders of Pregnancy; Preeclampsia; Gestational Hypertension
Keywords: Hypertensive disorders of pregnancy; Atorvastatin treatment; Pregnancy; Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced | interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: a double-blinded randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither participants, providers, investigators or outcome assessors will know to which of these groups participants are assigned. In case of an emergency, however, the study doctor can get this information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 10 mg Atorvastatin (Active Comparator): Atorvastatin 10 mg daily for 3 months
  Interventions: Drug: Atorvastatin 10 mg
- Placebo (Placebo Comparator): Identical appearing placebo for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin 10 mg — Participants will be assigned to 10 mg Atorvastatin
  Arms: 10 mg Atorvastatin
Drug: Placebo — Participants will be assigned to identical appearing placebo
  Arms: Placebo

SUMMARY:
The objective is to conduct a double-blinded randomized controlled trial of atorvastatin vs. placebo among postpartum individuals with hypertensive disorders of pregnancy, to improve cardiovascular risk score postpartum. For this, 76 individuals with hypertensive disorders of pregnancy (HDP) will be randomized to atorvastatin 10mg or placebo, which will be started in the postpartum period after cessation of breast feeding and continued for 3 months.

DETAILED DESCRIPTION:
Individuals will be followed for up to 1 year to address the following specific aims:

Specific Aim 1: To determine if among individuals diagnosed with hypertensive disorders of pregnancy (HDP), the use of atorvastatin 10 mg daily initiated in the postpartum period following cessation of breastfeeding and continued for 3 months, lowers cardiovascular risk, as measured by the Framingham Risk Score for Cardiovascular Disease (30 year risk, primary outcome) and cardiovascular risk prediction model (PREVENT, secondary outcome) compared with placebo; and if the benefit will persist for at least 3-6 months following discontinuation of atorvastatin treatment.

Specific Aim 2: To determine if among individuals diagnosed with HDP the use of atorvastatin 10 mg daily initiated in the postpartum period following cessation of breastfeeding and continued for 3 months lowers the frequency of metabolic syndrome, improves lipid levels, and reduces inflammatory markers compared with placebo; and if this benefit will persist for at least 3-6 months following discontinuation of atorvastatin treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Postpartum
2. ≥ 20 years old with the ability to give informed consent
3. Diagnosis of gestational hypertension, preeclampsia prior to delivery admission, or diagnosed with preeclampsia during delivery admission, as determined by clinical team using the American College of Obstetricians and Gynecologists (ACOG) criteria.
4. English speaking

Exclusion Criteria:

1. Individuals who were prescribed an 3-hydroxy-3 methyl-glutaryl coenzyme A (HMG-CoA) reductase inhibitor prior to or during pregnancy,
2. Known familial hypercholesterolemia or pre-existing hyperlipidemia, specifically Low-density Lipoprotein (LDL) >190 prior to pregnancy or diagnosis of hyperlipidemia with prescription of HMG-CoA reductase inhibitor prior to delivery,
3. Plan to breastfeed for >= 6 months,
4. Plan for pregnancy conception in the next 6 months,
5. Incarcerated individuals,
6. Hypertensive diagnosis thought to be secondary to fetal condition,
7. Contraindications to HMG-CoA reductase inhibitor therapy or known hypersensitivity to atorvastatin or any component,
8. Active liver disease (acute hepatitis, chronic active hepatitis, unexplained persistent transaminitis (at least twice upper limit of normal serum transaminases)),
9. History of rhabdomyolysis or myopathy,
10. Human Immunodeficiency Virus (HIV) positivity, due to potential interactions between atorvastatin and HIV protease inhibitors,
11. History of solid organ transplant, due to potential interactions between atorvastatin and immunosuppressants
12. Active cancer, or
13. Current use of medications with potential drug interactions, namely cyclosporine, clarithromycin, itraconazole, HIV protease inhibitors, rifampin, and digoxin.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 76 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
The 30-year Framingham Risk Score for Cardiovascular Disease | After 3 months of study treatment, up to 9 months after enrollment
  Predicts 0-100% risk of "hard" CVD events (coronary death, myocardial infarction, stroke) based on sex, systolic blood pressure, antihypertensive treatment, total and high-density lipoprotein cholesterol, smoking, and diabetes mellitus. A higher number reflects a greater risk of adverse CVD events, whereas a lower number reflects lower risk.

SECONDARY OUTCOMES:
Drug Use and Side Effects | From randomization until 6 months after stopping to use the study drug, up to 9 months
  Individuals will be contacted monthly via phone call to assess drug tolerability and use using a survey, which reviews any adverse events or concerns related to use of the study drug.
Framingham Risk Score for Cardiovascular Disease 3-6 months following medication cessation | Anytime after 3-6 months of stopping to use the study drug, up to 9 months from randomization
  Enrolled individuals will be contacted via telephone at 3-6 months after they complete medication use and will be invited to a visit for a Framingham Risk Score calculation. The Framingham Risk Score predicts 0-100% risk of CVD events, with a higher number reflecting a greater risk of adverse CVD events, whereas a lower number reflects lower risk.
PREVENT (AHA Predicting Risk of CVD Events) score | From randomization until 6 months after stopping to use the study drug, up to 9 months
  A glomerular filtration rate will be calculated for each enrolled individual upon enrollment and at the additional biospecimen visits in order to enable calculation of the PREVENT score.
Rates of primary care provider (PCP) visits within 9-12 months of delivery | From randomization until 6 months after stopping to use the study drug, up to 12 months from delivery
  Enrolled individuals will undergo a telephone survey at 9-12 months postpartum, assessing whether they have attended a visit with a primary care provider (internal medicine, family medicine or primary care nurse practitioner), and for what reason, since the time of their delivery
Waist circumference | From randomization until 6 months after stopping to use the study drug, up to 9 months
  Waist circumference in centimeters will be measured at the study visits to help identify those with metabolic syndrome (circumference of 88 cm or more).
Fasting glucose | From randomization until 6 months after stopping to use the study drug, up to 9 months
  Fasting glucose levels will be measured at the study visits to help identify those with metabolic syndrome (fasting glucose above or equal to 100 mg/dL).
Number of individuals diagnosed with metabolic syndrome | From randomization until 6 months after stopping to use the study drug, up to 9 months
  The presence of metabolic syndrome will be defined as 3 or more of the following, which are also listed as individual outcomes: waist circumference greater or equal to 88 cm, triglycerides greater or equal to 150 mg/dL, HDL cholesterol <50 mg/dL, blood pressure greater or equal to 130/85, and fasting glucose greater or equal to 100 mg/dL.
Lipid levels | From randomization until 6 months after stopping to use the study drug, up to 9 months
  Serum testing for total cholesterol, low-density lipoprotein cholesterol, very low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, and triglycerides
Hypertension diagnosis & need for antihypertensive therapy | From randomization until 6 months after stopping to use the study drug, up to 9 months
  Blood pressure will be measured at the study visits to identify new development of hypertension; enrolled individuals will be asked if they have started medication for hypertension
Diabetes diagnosis & need for anti-glycemic therapy | From randomization until 6 months after stopping to use the study drug, up to 9 months
  Hemoglobin A1C will be measured at the study visits to identify new development of diabetes mellitus (HbA1C > 6.5%) and individuals will be asked if they have started anti-glycemic medication
Systolic blood pressure | From randomization until 6 months after stopping to use the study drug, up to 9 months
Estimated glomerular filtration rate | From randomization until 6 months after stopping to use the study drug, up to 9 months
High-sensitivity C-reactive protein (Hs-CRP) level | From randomization until 6 months after stopping to use the study drug, up to 9 months
Lipoprotein (a) level | From randomization until 6 months after stopping to use the study drug, up to 9 months
Apolipoprotein (b) level | From randomization until 6 months after stopping to use the study drug, up to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Tracy C Bank, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center OB/GYN Maternal and Fetal Medicine, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No